CLINICAL TRIAL: NCT04411433
Title: An Open-Label, Multicenter, Parallel-Group, Randomized, Phase III Study to Evaluate the Efficacy and Safety of Hydroxychloroquine and Favipiravir in the Treatment of Mild to Moderate COVID-19
Brief Title: Efficacy and Safety of Hydroxychloroquine and Favipiravir in the Treatment of Mild to Moderate COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ministry of Health, Turkey (Other Government)
Collaborators: Hacettepe University (Other); Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other); Umraniye Education and Research Hospital (Other Government); SB Istanbul Education and Research Hospital (Other); Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other); Tepecik Training and Research Hospital (Other); Istanbul University - Cerrahpasa (Other); Ankara University (Other); Ankara City Hospital Bilkent (Other); Ankara Training and Research Hospital (Other); Ege University Hospital (Application and Research Center) (Unknown); Kocaeli Derince Education and Research Hospital (Other); Istanbul University (Other); Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Prof. Ates KARA, MD, Prof., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVID-19-FAV
Record Dates: First submitted 2020-05-23; First posted 2020-06-02 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Sars-CoV2; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — favipiravir; Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Intervention Model Description: This is an open-label, multicenter, parallel-group, randomized, phase III trial that evaluates the efficacy and safety of hydroxychloroquine and favipiravir in the treatment of patients with possible or confirmed COVID-19 observed within the last 5 days. 1000 patients will be randomized in 2:1:2:2:2:1 ratio and divided into six groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Favipiravir (3200 mg + 1200 mg) (Experimental): Dosage and method of administration: in a regimen of 2x1600 mg (oral) loading dose on day-1 followed by 1200 mg maintenance dose (2x600 mg, 2 times daily) on day-2 to day-5 (5 days in total).
  The treatment duration may be extended up to 14 days with the evaluation of principle investigator.
  Interventions: Drug: Favipiravir (3200 mg + 1200 mg)
- Favipiravir (3600 mg + 1600 mg) (Experimental): Dosage and method of administration: in a regimen of 2x1800 mg (oral) loading dose on day-1 followed by 1600 mg maintenance dose (2x800 mg, 2 times daily) on day-2 to day-5 (5 days in total).
  The treatment duration may be extended up to 14 days with the evaluation of principle investigator.
  Interventions: Drug: Favipiravir (3600 mg + 1600 mg)
- Favipiravir combined with Hydroxychloroquine (Experimental): Hydroxychloroquine Dosage and method of administration: in a regimen of 2x400 mg (oral) loading dose on day-1 followed by 400 mg maintenance dose (2x200 mg oral, 2 times daily) on day-2 to day-5 (5 days in total).
  Favipiravir Dosage and method of administration: in a regimen of 2x1600 mg (oral) loading dose on day-1 followed by 1200 mg maintenance dose (2x600 mg, 2 times daily) on day-2 to day-5 (5 days in total). The treatment duration may be extended up to 14 days with the evaluation of principle investigator.
  Interventions: Drug: Favipiravir (3200 mg + 1200 mg) combined with Hydroxychloroquine
- Favipiravir combined with Azithromycin (Experimental): Azithromycin Dosage and method of administration: in a regimen of 1x500 mg (oral) loading dose on day-1 followed by 250 mg maintenance dose (oral daily) on day-2 to day-5 (5 days in total).
  Favipiravir Dosage and method of administration: in a regimen of 2x1600 mg (oral) loading dose on day-1 followed by 1200 mg maintenance dose (2x600 mg, 2 times daily) on day-2 to day-5 (5 days in total). The treatment duration may be extended up to 14 days with the evaluation of principle investigator.
  Interventions: Drug: Favipiravir (3200 mg + 1200 mg) combined with Azithromycin
- Hydroxychloroquine (Active Comparator): Dosage and method of administration for patients with mild possible or confirmed COVID-19 pneumonia (no severe pneumonia symptoms): in a regimen of 2x400 mg (oral) loading dose on day-1 followed by 400 mg maintenance dose (200 mg oral 2 times daily) on day-2 to day-5 (5 days in total).
  Dosage and method of administration for patients with uncomplicated possible or confirmed COVID-19: in a regimen of 400 mg (200 mg oral 2 times daily) throughout 5 days (5 days in total).
  Interventions: Drug: Hydroxychloroquine
- Hydroxychloroquine combined with Azithromycin (Active Comparator): Hydroxychloroquine Dosage and method of administration for patients with mild possible or confirmed COVID-19 pneumonia (no severe pneumonia symptoms): in a regimen of 2x400 mg (oral) loading dose on day-1 followed by 400 mg maintenance dose (2x200 mg oral, 2 times daily) on day-2 to day-5 (5 days in total).
  Hydroxychloroquine Dosage and method of administration for patients with uncomplicated possible or confirmed COVID-19: in a regimen of 400 mg (2x200 mg oral, 2 times daily) throughout 5 days (5 days in total).
  Azithromycin Dosage and method of administration: in a regimen of 1x500 mg (oral) loading dose on day-1 followed by 250 mg maintenance dose (oral daily) on day-2 to day-5 (5 days in total).
  Interventions: Drug: Hydroxychloroquine combined with Azithromycin

INTERVENTIONS:
Drug: Favipiravir (3200 mg + 1200 mg) — Dosage and method of administration: in a regimen of 2x1600 mg (oral) loading dose on day-1 followed by 1200 mg maintenance dose (2x600 mg, 2 times daily) on day-2 to day-5 (5 days in total).
  The treatment duration may be extended up to 14 days with the evaluation of principle investigator.
  Arms: Favipiravir (3200 mg + 1200 mg)
Drug: Favipiravir (3600 mg + 1600 mg) — Drug: Favipiravir (3600 mg + 1600 mg) Dosage and method of administration: in a regimen of 2x1800 mg (oral) loading dose on day-1 followed by 1600 mg maintenance dose (2x800 mg, 2 times daily) on day-2 to day-5 (5 days in total).
  The treatment duration may be extended up to 14 days with the evaluation of principle investigator.
  Arms: Favipiravir (3600 mg + 1600 mg)
Drug: Favipiravir (3200 mg + 1200 mg) combined with Hydroxychloroquine — Hydroxychloroquine Dosage and method of administration: in a regimen of 2x400 mg (oral) loading dose on day-1 followed by 400 mg maintenance dose (2x200 mg oral, 2 times daily) on day-2 to day-5 (5 days in total).
  Favipiravir Dosage and method of administration: in a regimen of 2x1600 mg (oral) loading dose on day-1 followed by 1200 mg maintenance dose (2x600 mg, 2 times daily) on day-2 to day-5 (5 days in total). The treatment duration may be extended up to 14 days with the evaluation of principle investigator.
  Arms: Favipiravir combined with Hydroxychloroquine
Drug: Favipiravir (3200 mg + 1200 mg) combined with Azithromycin — Azithromycin Dosage and method of administration: in a regimen of 1x500 mg (oral) loading dose on day-1 followed by 250 mg maintenance dose (oral daily) on day-2 to day-5 (5 days in total).
  Favipiravir Favipiravir Dosage and method of administration: in a regimen of 2x1600 mg (oral) loading dose on day-1 followed by 1200 mg maintenance dose (2x600 mg, 2 times daily) on day-2 to day-5 (5 days in total). The treatment duration may be extended up to 14 days with the evaluation of principle investigator.
  Arms: Favipiravir combined with Azithromycin
Drug: Hydroxychloroquine — Dosage and method of administration for patients with mild possible or confirmed COVID-19 pneumonia (no severe pneumonia symptoms): in a regimen of 2x400 mg (oral) loading dose on day-1 followed by 400 mg maintenance dose (200 mg oral 2 times daily) on day-2 to day-5 (5 days in total).
  Dosage and method of administration for patients with uncomplicated possible or confirmed COVID-19: in a regimen of 400 mg (200 mg oral 2 times daily) throughout 5 days (5 days in total).
  Arms: Hydroxychloroquine
Drug: Hydroxychloroquine combined with Azithromycin — Drug: Hydroxychloroquine combined with Azithromycin Hydroxychloroquine Dosage and method of administration for patients with mild possible or confirmed COVID-19 pneumonia (no severe pneumonia symptoms): in a regimen of 2x400 mg (oral) loading dose on day-1 followed by 400 mg maintenance dose (2x200 mg oral, 2 times daily) on day-2 to day-5 (5 days in total).
  Hydroxychloroquine Dosage and method of administration for patients with uncomplicated possible or confirmed COVID-19: in a regimen of 400 mg (2x200 mg oral, 2 times daily) throughout 5 days (5 days in total).
  Azithromycin Dosage and method of administration: in a regimen of 1x500 mg (oral) loading dose on day-1 followed by 250 mg maintenance dose (oral daily) on day-2 to day-5 (5 days in total).
  Arms: Hydroxychloroquine combined with Azithromycin

SUMMARY:
This is an open-label, multicenter, parallel-group, randomized, phase III trial that evaluates the efficacy and safety of hydroxychloroquine and favipiravir in the treatment of patients with possible or confirmed COVID-19 observed within the last 5 days. 1000 patients will be randomized in 2:1:2:2:2:1 ratio and divided into six groups.

DETAILED DESCRIPTION:
The clinical picture of 2019-nCoV disease is in a broad spectrum, which includes asymptomatic infection, a mild upper respiratory tract infection, respiratory failure, and even severe viral pneumonia with death. Although the mortality rate is not yet clear, the reported case-fatality risk was 11-14% during the initial studies which included patients with severe disease. The overall case fatality rate was reported as approximately 2%. In addition, most cases have resulted in a pneumonia requiring supplemental oxygen therapy and ventilator support. The alarming levels of spread and severity of COVID-19 caused a global emergency and this outbreak has been characterized as a pandemic by the World Health Organization (WHO).

The investigational product Favipiravir is an antiviral drug against RNA viruses and has been stated as effective for the treatment of COVID-19, first emerged from China, in various clinical studies. In February 2020, Favipiravir was used for the clinical treatment of COVID-19, has been shown to be more effective than the lopinavir / ritonavir combination in 80 people. In recent researches, the drug favipiravir is suggested that it may induce recovery in a short time in patients with COVID-19-mild type and decrease the treatment duration from 11 days to 4 days.

The investigational product hydroxychloroquine sulfate is a 4- aminoquinoline derivative and widely used for the treatment of many rheumatic diseases such as rheumatoid arthritis and systemic lupus erythematosus in addition to its antimalarial effects. In vitro studies reported that hydroxychloroquine sulfate may be effective against many viruses, including SARS-CoV-2 in many in vitro experiments. Additionally, preliminary results of limited number of studies have been revealed that hydroxychloroquine sulfate reduces virus load and induces improvement in patients with COVID-19. This agent has been also suggested to be used in COVID-19 prophylaxis.

Until now, there is no official report on whether hydroxychloroquine combined with favipiravir show clinical activity against the new coronavirus, COVID-19, in Turkey. The main purpose of this study is to evaluate the efficacy and safety of hydroxychloroquine and favipiravir in the treatment of Turkey population with COVID-19.

This study designed as an open-label, multicenter, parallel-group, randomized, phase III clinical drug trial.

A total of 1000 subjects aged between 18 to 70 years with symptoms and complaints consistent with possible or confirmed COVID-19 observed within the last 5 days and meet all eligibility criteria will participate in the study.

This study will be conducted in 14 sites.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 to 70 years,
* Patients with symptoms and complaints consistent with possible or confirmed COVID- 19 observed within the last 5 days,
* Patients with uncomplicated possible or confirmed COVID-19:

  1. Symptoms such as fever, muscle aches, joint pain, cough, sore throat, nasal congestion, however no respiratory distress, no tachypnea or no SpO2 < 93%,
  2. Chest imaging (X-ray or CT chest) documented as normal
* Patients with mild possible or confirmed COVID-19 pneumonia (no severe pneumonia symptoms):

  1. Symptoms such as fever, muscle aches, joint pain, cough, sore throat, nasal congestion, as well as respiratory rate <30/min and SpO2 above 93% on room air,
  2. Chest imaging (X-ray or CT chest)-documented mild pneumonia symptoms
* Patients who were decided to isolate and treat because of COVID-19 in the hospital,
* Patients who have not been involved in any other interventional studies.

Exclusion Criteria:

* Patients considered as inappropriate for this study for any reason like noncompliance by the researcher,
* Patients with persisting refractory nausea, vomiting, chronic diarrhoea or chronic gastrointestinal disorders, inability to swallow the study drug which may affect adequate absorption,
* Patients with chronic liver disease: alanine aminotransferase (ALT)/aspartate aminotransferase (AST) elevated over 5 times the upper limit of normal (ULN),
* Patients with gout or hyperuricemia (above the ULN),
* Patients with severe pneumonia symptoms,
* Patients with known allergy to Favipiravir or for substances used in the study,
* Patients did not receive specific antiviral drugs such as lopinavir/ritonavir, ribavirin, arbidol, chloroquine phosphate, hydroxychloroquine, and monoclonal antibodies within one week before admission.
* Patients with known chronic renal impairment/failure [creatinine clearance (CcCl) <30 mL/min],
* Pregnant and lactating women
* Patients undergoing cardiac ablation therapy
* Patients using antiarrhythmic drugs
* Patients actively receiving chemotherapy
* Acute immunosuppressed patients
* Patients undergoing psychosis therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1008 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Time to recovery (discharge) | 14 days
  The evaluation of recovery (discharge) period until 14th day after administration.
Decrease in viral load | 14 days
  The evaluation of decrease in viral load until 14th day after administration.

SECONDARY OUTCOMES:
Adverse Event (AE), Serious Adverse Event (SAE) and discontinuation of treatment | 14 days
  Number/characteristics of Adverse Event (AE), Serious Adverse Event (SAE) and discontinuation of treatment due to study drug from baseline until the end of study
Frequency of occurrence of lymphopenia from baseline | 14 days
  Clinical evaluation of occurrence of lymphopenia from baseline until the end of study.
Frequency of occurrence of thrombocytopenia from baseline | 14 days
  Clinical evaluation of occurrence of thrombocytopenia from baseline until the end of study.
Changes in alanine aminotransferase (ALT) levels from baseline | 14 days
  Clinical evaluation of ALT levels from baseline until the end of study.
Changes in aspartate aminotransferase (AST) levels from baseline | 14 days
  Clinical evaluation of AST levels from baseline until the end of study.
Changes in C-reactive protein (CRP) levels from baseline | 14 days
  Clinical evaluation of CRP levels from baseline until the end of study.
Changes in level of D-dimer levels from baseline | 14 days
  Clinical evaluation of D-dimer levels from baseline until the end of study.
Changes in prothrombin time (PT) values from baseline | 14 days
  Clinical evaluation of PT values for blood to coagulate from baseline until the end of study.
Changes in partial thromboplastin time (PTT) values from baseline | 14 days
  Clinical evaluation of PTT values for blood to coagulate from baseline until the end of study.
Changes in blood pressure from baseline | 14 days
  Clinical evaluation of systolic and diastolic blood pressure levels from baseline until the end of study.
Changes in respiratory rate from baseline | 14 days
  Clinical evaluation of respiratory rate levels from baseline until the end of study.
Changes in pulse oxymetry from baseline | 14 days
  Clinical evaluation of pulse oxymetry levels from baseline until the end of study.
Changes in fever from baseline | 14 days
  Clinical evaluation of changes in fever from baseline until the end of study.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, School of Medicine, Ankara, Turkey (Türkiye)